CLINICAL TRIAL: NCT06189872
Title: Radiographic Migration Analysis of the ATTUNE Cementless CR Fixed-Bearing Total Knee Replacement: A Multi-Center, Non-Controlled, Prospective Study
Brief Title: Radiographic Migration Analysis of the ATTUNE Cementless CR Fixed-Bearing Total Knee Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATTUNE2024
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Attune Cementless, Fixed Bearing, Cruciate Retaining TKA System (Other): Attune Cruciate Retaining TKA System
  Interventions: Device: Attune Cementless

INTERVENTIONS:
Device: Attune Cementless — * Attune AFFIXIUM Cementless Tibial Baseplate, Fixed Bearing
  * Attune POROCOAT Cementless Femoral Component, Cruciate Retaining
  * Attune AOX Antioxidant Polyethylene Tibial Insert, Cruciate Retaining
  * Attune AOX Patellar Button, Domed or Medialized Dome, Cemented or Cementless (surgeon preference for resurfacing)

SUMMARY:
This is a multi-centre, single cohort trial of patients undergoing cruciate-retaining total knee arthroplasty with the Attune Cementless, Fixed Bearing, Cruciate Retaining TKA System.

DETAILED DESCRIPTION:
All patients will undergo post-operative radiostereometric analysis (RSA) and computed tomography (CT) to quantify and characterize the in vivo migration pattern of the Attune AFFIXIUM Cementless Tibial Baseplate and the Attune POROCOAT Cementless Femoral Component up to 24 months. Patient health and functional outcomes will be recorded at pre- and post-operative intervals for all patients. Peri-operative adverse events and other clinical complications will be captured as encountered.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating primary total knee arthroplasty
* Patients aged 21 years or older
* Sufficient ligamentous function to warrant retention of the posterior cruciate ligament
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent

Exclusion Criteria:

* Active or prior infection of ipsilateral extremity
* Medical condition precluding major surgery
* Inflammatory arthropathy
* Posterior cruciate ligament (PCL) deficiency
* Major coronal plane deformity
* Conditions that are cautioned against or contraindicated, as listed in the product monograph and/or instruction for use
* Bone defects requiring augments, cones and/or stemmed implants

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Tibial baseplate stability | 6-12 months, 1-2 years post-operative
  Maximum total point motion (MTPM) migration between 6-12 months and 1-2 year post-operative (mm)

SECONDARY OUTCOMES:
Femoral component migration | Discharge, 6 Weeks, 6 Months, 1 Year and 2 Years
  To quantify and characterize femoral component migration up to 24 months after surgery
Tibial baseplate migration | Discharge, 6 Weeks, 6 Months, 1 Year and 2 Years
  To quantify and characterize tibial baseplate migration between weight-bearing and non-weight-bearing examinations at 24 months after surgery.
Equivalency between CT-RSA-measured migration and the gold-standard of RSA-measured migration | Discharge, 6 Weeks, 6 Months, 1 Year and 2 Years
  To assess equivalency between CT-RSA-measured migration and the gold-standard of RSA-measured migration for both tibial and femoral migration
European Quality of Life (EQ-5D-5L) | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  EQ5D consists of 5 subscales; Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety / depression. A health state score is obtained based on the responses from 1-5 in each subscale, from which a single index value is calculated representing patients' overall health state. EQ5D includes a so called EQ VAS score which is the patients' self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Oxford Knee Score | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  The Oxford Knee Score (OKS) is a patient self-administered 12-item questionnaire with each question having a Likaert-like response option. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance. The OKS measures pain and general activities of daily living.
Forgotten Joint Score (FJS) | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  The FJS total score range is 0-100, higher scores indicating the patient is able to forget the joint daily or lower degree of joint awareness.
Satisfaction VAS | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported pain severity as measured using the visual analogue scale (VAS) from 0 (Unsatisfied) - 100 (Completely satisfied)
Patient complications | Preoperative, 6 Weeks, 6 Months, 1 Year and 2 Years
  Evaluate the type and frequency of the complications/adverse events.
Linear depth (wear) on the tibial insert | Discharge, 6 Weeks, 6 Months, 1 Year and 2 Years
  To estimate linear depth (wear) on the tibial insert (experimental).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — Concordia Hospital
Locations (3):
- Canada (3):
  - Orthopaedic Innovation Centre, Winnipeg, Manitoba
  - Nova Scotia Health - Orthopedic, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario